CLINICAL TRIAL: NCT07068490
Title: Impact of Potassium Competitive Acid Blockers After Percutaneous Coronary Intervention for Efficacy and Safety Outcome: Target Trial Emulation Study.
Acronym: PCAB-PCI
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Associate Professor, Samsung Medical Center
Other Study IDs: PCAB_TTE
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: percutaeneous coronary intervention; dual antiplatelet therapy; gastrointestinal protection
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine use of P-CAB: All-comer patients with P-CAB
  Interventions: Drug: Routine use of P-CAB on DAPT
- Guideline-directed GI protection strategy: Use of PPI or not according to GI bleeding risk
  Interventions: Drug: Guideline Directed Medical Therapy

INTERVENTIONS:
Drug: Routine use of P-CAB on DAPT — This group received P-CAB with DAPT after PCI.
  Groups: Routine use of P-CAB
Drug: Guideline Directed Medical Therapy — This group received PPI or not with DAPT after PCI according to GI bleeding risk.
  Groups: Guideline-directed GI protection strategy

SUMMARY:
Despite the fact that potassium competitive acid blocker (P-CAB) has been developed for the treatment of gastric ulcer or gastroesophageal reflux disease, the efficacy and safety of P-CAB for the use of gastrointestinal (GI) protection in patients undergoing percutaneous coronary intervention (PCI) and maintaining dual antiplatelet therapy (DAPT) remains uncertain.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of routine P-CAB use in patients with coronary artery disease who underwent PCI and maintain DAPT, as compared to guideline-directed proton pump inhibitor (PPI) usage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent PCI
* Use of either clopidogrel, prasugrel, or ticagrelor in combination with aspirin
* No use of PCAB, PPI, or an H2-receptor within the past month

Exclusion Criteria:

* Patients with low GI bleeding risk are taken on PPI
* Patients with high GI bleeding risk do not take PPI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease who underwent PCI
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major GI bleeding | at 1 year
  Major GI bleeding requiring transfusion

SECONDARY OUTCOMES:
Clinically relevant GI bleeding | At 1 year
  Clinically relevant GI bleeding
Major adverse cardiac event | At 1 year
  A composite of cardiovascular death, myocardial infarction, and repeat revascularization
Cardiovascular death | At 1 year
  Cardiovascular death
Myocardial infarction | At 1 year
  Myocardial infarction
Repeat revascularization | At 1 year
  Repeat revascularization

CONTACTS AND LOCATIONS:
Overall Officials: KI HONG CHOI, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided